CLINICAL TRIAL: NCT04109560
Title: High Flow Nasal Oxygen Therapy in Chronic Obstructive Pulmonary Disease (COPD) Patients With Acute Hypercapnic Respiratory Failure (AHRF)
Brief Title: HFNC and Acute Hypercapnic Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Principal Investigator, Gustavo Plotnikow, Physical Therapist, Argentinian Intensive Care Society
Other Study IDs: Hi-VNI in AHRF
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: High Flow Oxygen Therapy; Acute Hypercapnic Respiratory Failure; COPD Exacerbation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High-flow nasal cannula (HFNC) enables delivering humidified gas at high-flow rates controlling the oxygen inspired fraction (FiO2). Its efficacy has been demonstrated in hypoxemic acute respiratory failure. However, little is known about its use in hypercapnic acute respiratory failure (ARF). Therefore, we aimed to evaluate the effect of using HFNC through "Precision Flow" equipment as first line of ventilatory support for COPD patients with hypercapnic acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to very severe COPD patients (GOLD 2 to 4) over 18 years old admitted to the ICU with hypercapnic ARF (PaCO2> 45 mmHg and respiratory acidosis [pH ≥7.30], with or without hypoxemia + one of the following: Respiratory Rate ≥25 cycles per minute, intercostal and / or supraclavicular recruitment, or thoraco-abdominal synchrony, no prior use of NIV)

Exclusion Criteria:

* Patients less than 18 years old
* Mild COPD patients
* Absence of hypercapnia
* Kelly M Score > 3
* Haemodynamic instability (despite fluid resuscitation)
* NIV or Invasive Mechanical Ventilation (IMV) (Need to use previously to HFNC)
* Contraindications to implement high-flow oxygen therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to very severe COPD patients (GOLD 2 to 4) admitted to the ICU with acute hypercapnic respiratory failure
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Need for non-invasive ventilation | From inclussion study date until the first day of noninvasive ventilation use documented, after high flow oxygen therapy use or death date from any cause, whichever came first, assessed up to 4 weeks.
  The need and causes for non-invasive ventilation will be recorded in the all study period.
Need for endotracheal intubation | From inclussion study date until the first day of endotracheal intubation documented, after high flow oxygen therapy use or death date from any cause, whichever came first, assessed up to 4 weeks.
  The need and causes for endotracheal intubation will be recorded in the all study period.

SECONDARY OUTCOMES:
Gas Exchange | Arterial blood gases will be recorded 1, 24 hours and every 24 hours after enrollment
  pH will be recorded
Gas Exchange | Arterial blood gases will be recorded 1, 24 hours and every 24 hours after enrollment
  PaCO2 in milimeters of mercury (mmHg) will be recorded
Gas Exchange | Arterial blood gases will be recorded 1, 24 hours and every 24 hours after enrollment
  PaO2 in milimeters of mercury (mmHg) will be recorded
Respiratory variables | Respiratory variables will be recorded at 1, 2, 3, 6, 12, 24 hours and every 24 hours after enrollment
  Respiratory rate in numbers of breaths per minute (bpm) will be recorded
Respiratory variables | Respiratory variables will be recorded at 1, 2, 3, 6, 12, 24 hours and every 24 hours after enrollment
  Accessory muscular use (intercostal or supraclavicular) by "YES or NO" will be recorded
Respiratory variables | Respiratory variables will be recorded at 1, 2, 3, 6, 12, 24 hours and every 24 hours after enrollment
  Thoraco-abdominal asynchrony by "YES or NO" will be recorded
Patient's discomfort | Patient's discomfort will be recorded at 1, 2, 3, 6, 12, 24 hours and every 24 hours after enrollment
  Discomfort related to the high flow oxygen therapy and related to the degree of humidification will be assessed by using a numerical rating scale from 1 (no discomfort) to 5 (maximum imaginable discomfort). Patients will be asked to rate their discomfort with the used device and discomfort symptoms will be determined for the dryness of the delivered oxygen (dryness of the mouth, throat, nose, difficulty to swallow and throat pain).

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo A Plotnikow, Study Director — Sanatorio Anchorena Recoleta; Mariano Setten, Principal Investigator — Centro de Educación Médica e Investigaciones Clínicas "Norberto Quirno" (CEMIC); Norberto Tiribelli, Principal Investigator — Complejo Médico Policial Churruca-Visca; Sebastian Fredes, Principal Investigator — Sanatorio de la Trinidad Mitre; Matias Accoce, Principal Investigator — Sanatorio Anchorena San Martín
Locations (1):
- Sanatorio Anchorena, CABA, Argentina